CLINICAL TRIAL: NCT01468207
Title: A Phase 3 Multicenter Study of the Safety and Efficacy of Adalimumab in Subjects With Moderate to Severe Hidradenitis Suppurativa - PIONEER I
Brief Title: Efficacy and Safety Study of Adalimumab in Treatment of Hidradenitis Suppurativa
Acronym: PIONEER I
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M11-313; 2011-003400-20 (EudraCT Number)
Record Dates: First submitted 2011-11-07; First posted 2011-11-09 (Estimated); Results first posted 2015-10-28 (Estimated); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Hidradenitis Suppurativa (HS)
Keywords: acne; psoriasis; hidradenitis suppurativa; TNF; HS; PIONEER I; acne inversa; boil; placebo controlled; Double blind; adalimumab
MeSH Terms: conditions — Hidradenitis Suppurativa; Acne Vulgaris; Psoriasis; Furunculosis | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Placebo (Placebo Comparator): Placebo for 12 weeks.
  Interventions: Biological: placebo
- Adalimumab Every Week (EW) (Experimental): Adalimumab ew for 12 weeks (160 mg at Week 0; 80 mg at Week 2; and 40 mg ew from Week 4 to Week 12).
  Interventions: Biological: adalimumab
- Placebo/Adalimumab Every Week (EW) (Experimental): Participants randomized to receive placebo in Period 1 received adalimumab 160 mg at Week 12, 80 mg at Week 14, and 40 mg ew from Week 16 to Week 35 in Period 2 (up to 24 weeks).
  Interventions: Biological: adalimumab; Biological: placebo
- Adalimumab Every Week (EW)/Placebo (Experimental): Participants randomized to receive adalimumab ew in Period 1 were re-randomized to receive placebo ew from Week 12 to Week 35 in Period 2 (up to 24 weeks).
  Interventions: Biological: adalimumab; Biological: placebo
- Adalimumab Every Week (EW)/ Adalimumab Every Other Week (EOW) (Experimental): Participants randomized to receive adalimumab ew in Period 1 were re-randomized to receive adalimumab 40 mg eow from Week 12 to Week 35 in Period 2; placebo injections were administered eow from Week 13 to Week 35 (up to 24 weeks).
  Interventions: Biological: adalimumab
- Adalimumab Every Week (EW)/Adalimumab Every Week (EW) (Experimental): Participants randomized to receive adalimumab ew in Period 1 were re-randomized to receive 40 mg adalimumab ew from Week 12 to Week 35 in Period 2 (up to 24 weeks).
  Interventions: Biological: adalimumab

INTERVENTIONS:
Biological: adalimumab — Adalimumab pre-filled syringe, administered by subcutaneous injection
  Other Names: Humira
  Arms: Adalimumab Every Week (EW); Adalimumab Every Week (EW)/ Adalimumab Every Other Week (EOW); Adalimumab Every Week (EW)/Adalimumab Every Week (EW); Adalimumab Every Week (EW)/Placebo; Placebo/Adalimumab Every Week (EW)
Biological: placebo — Placebo pre-filled syringe, administered by subcutaneous injection
  Arms: Adalimumab Every Week (EW)/Placebo; Placebo; Placebo/Adalimumab Every Week (EW)

SUMMARY:
A study to evaluate the safety and efficacy of treatment with adalimumab in adults with moderate to severe hidradenitis suppurativa (HS).

DETAILED DESCRIPTION:
The clinical trial identifier is PIONEER I. The purpose of this study is to evaluate the safety of adalimumab and to determine how well it works in the treatment of adults with moderate to severe HS. HS is a chronic skin disease that creates red, swollen, painful bumps which can break open to combine and form tunnels in the skin and scars. Sometimes these bumps can heal themselves quickly and sometimes they will become much worse and create sores that heal with multiple combined scars, or areas that do not heal. In this study, approximately 300 adults will be enrolled at treatment centers worldwide. Subject participation in this study will be up to 50 weeks. There will be a screening period, which will last from 7 to 30 days, and a study treatment period of up to 36 weeks. Study visits occur at Screening, Baseline, and Weeks 2, 4, 8, 12, 14, 16, 20, 24, 28, 32 and 36 (or sooner if subject leaves the study before Week 36). The study is divided into two treatment periods. The first period (Period A) will last 12 weeks and the second period (Period B) will last up to 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adults must have a diagnosis of HS for at least 1 year prior to Baseline.
* HS lesions must be present in at least two distinct anatomical areas, one of which must be at least Hurley Stage II or Hurley Stage III.
* Subject must have stable HS for at least 60 days prior to Screening visit and at Baseline visit.
* Subject must have experienced an inadequate response to at least a 90-day treatment of oral antibiotics for treatment of HS.
* Subject must have a total AN count of greater than or equal to 3 at baseline.

Exclusion Criteria:

* Subject was previously treated with adalimumab or another anti-tumor necrosis factor (anti-TNF) therapy (e.g., infliximab or etanercept).
* Subject received any oral antibiotic treatment for HS within 28 days prior to Baseline.
* Subject received oral concomitant analgesics (including opioids) for HS-related pain within 14 days prior to Baseline visit.
* If entering the study on concomitant oral analgesics for non-HS related pain:

  * Subject on opioid analgesics within 14 days prior to Baseline visit;
  * Subject not on a stable dose of non-opioid oral analgesics for at least 14 days prior to the Baseline visit ("as needed" is not considered a stable dose).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2011-11; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Williams, MD, Study Chair — AbbVie

REFERENCES:
- [Result] Kimball AB, Okun MM, Williams DA, Gottlieb AB, Papp KA, Zouboulis CC, Armstrong AW, Kerdel F, Gold MH, Forman SB, Korman NJ, Giamarellos-Bourboulis EJ, Crowley JJ, Lynde C, Reguiai Z, Prens EP, Alwawi E, Mostafa NM, Pinsky B, Sundaram M, Gu Y, Carlson DM, Jemec GB. Two Phase 3 Trials of Adalimumab for Hidradenitis Suppurativa. N Engl J Med. 2016 Aug 4;375(5):422-34. doi: 10.1056/NEJMoa1504370. PMID 27518661
- [Derived] Kearney N, Chen X, Bi Y, Hew K, Smith KM, Kirby B. Treatment of hidradenitis suppurativa with adalimumab in the PIONEER I and II randomized controlled trials reduced indices of systemic inflammation, recognized risk factors for cardiovascular disease. Clin Exp Dermatol. 2025 Jan 27;50(2):339-347. doi: 10.1093/ced/llae324. PMID 39141589
- [Derived] Ryan C, Sobell JM, Leonardi CL, Lynde CW, Karunaratne M, Valdecantos WC, Hendrickson BA. Safety of Adalimumab Dosed Every Week and Every Other Week: Focus on Patients with Hidradenitis Suppurativa or Psoriasis. Am J Clin Dermatol. 2018 Jun;19(3):437-447. doi: 10.1007/s40257-017-0341-6. PMID 29380251
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants ≥ 18 years of age with HS for at least 1 year prior to Baseline and HS lesions present in at least 2 distinct anatomical areas (one of which must be at least Hurley Stage II or III) who had experienced inadequate response to ≥ 90 day treatment of oral antibiotics for HS were eligible for enrolment in the study.
Period: Treatment Period 1
Arm/Group | Placebo | Adalimumab Every Week (EW) | Placebo/Adalimumab Every Week (EW) | Adalimumab Every Week (EW)/Placebo | Adalimumab Every Week (EW)/ Adalimumab Every Other Week (EOW) | Adalimumab Every Week (EW)/Adalimumab Every Week (EW)
Started | 154 | 153 | 0 | 0 | 0 | 0
Received Study Drug | 152 | 153 | 0 | 0 | 0 | 0
Completed | 145 | 145 | 0 | 0 | 0 | 0
Not Completed | 9 | 8 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 5 | 4 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 2 | 0 | 0 | 0 | 0
Period: Treatment Period 2
Arm/Group | Placebo | Adalimumab Every Week (EW) | Placebo/Adalimumab Every Week (EW) | Adalimumab Every Week (EW)/Placebo | Adalimumab Every Week (EW)/ Adalimumab Every Other Week (EOW) | Adalimumab Every Week (EW)/Adalimumab Every Week (EW)
Started | 0 | 0 | 145 | 49 | 48 | 48
Completed | 0 | 0 | 93 | 22 | 27 | 28
Not Completed | 0 | 0 | 52 | 27 | 21 | 20
Not completed — Adverse Event | 0 | 0 | 6 | 1 | 2 | 1
Not completed — Lack of Efficacy | 0 | 0 | 1 | 1 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 5 | 0 | 0 | 2
Not completed — Loss/abscence of response (per protocol) | 0 | 0 | 30 | 23 | 18 | 13
Not completed — Lost to Follow-up | 0 | 0 | 5 | 1 | 0 | 0
Not completed — Other | 0 | 0 | 5 | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Adalimumab Every Week (EW) | Total
Number analyzed (Participants) | 154 | 153 | 307
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (11.33) | 36.2 (10.83) | 37.0 (11.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 91 | 196
  Male | 49 | 62 | 111

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Hidradenitis Suppurativa Clinical Response (HiSCR) at Week 12
Description: HiSCR was defined as at least a 50% reduction in abscess and inflammatory nodule (AN) count with no increase in abscess count and no increase in draining fistula count at Week 12 relative to Baseline. Data are presented for all participants and by baseline Hurley Stage (Stage 1: Abscess formation, single or multiple, without sinus tracts and scarring; Stage II: One or more widely separated recurrent abscesses with tract formation and scars. A participant with at least 1 anatomic region with Hurley Stage II disease and with no anatomic regions with Hurley Stage III disease was classified as Hurley Stage II; and Stage III: Multiple interconnected tracts and abscesses across the entire area, with diffuse or near diffuse involvement. A participant with at least 1 anatomic region with Hurley Stage III disease was classified as Hurley Stage III). Non-responder imputation (NRI): Participants with missing data were considered non-responders.
Time Frame: Baseline (Week 0) up to Week 12
Population: The intention-to-treat (ITT) population, defined as all participants who were randomized at Baseline (Week 0), was analyzed overall and by baseline Hurley Stage
Measure: Number; unit: percentage of participants
Groups:
- Placebo - Baseline Hurley Stage II: Participants with baseline Hurley Stage II randomized to receive placebo every week (ew) for 12 weeks.
- Placebo - Baseline Hurley Stage III: Participants with baseline Hurley Stage III randomized to receive placebo every week (ew) for 12 weeks.
- Adalimumab Every Week (EW) - Baseline Hurley Stage II: Participants with baseline Hurley Stage II randomized to receive adalimumab ew 160 mg at Week 12, 80 mg at Week 14, and 40 mg ew from Week 16 to 35 (up to 24 weeks).
- Adalimumab Every Week (ew) - Baseline Hurley Stage III: Participants with baseline Hurley Stage III randomized to receive adalimumab ew 160 mg at Week 12, 80 mg at Week 14, and 40 mg ew from Week 16 to 35 (up to 24 weeks).
Arm/Group | Placebo | Adalimumab Every Week (EW) | Placebo - Baseline Hurley Stage II | Placebo - Baseline Hurley Stage III | Adalimumab Every Week (EW) - Baseline Hurley Stage II | Adalimumab Every Week (ew) - Baseline Hurley Stage III
Number analyzed (Participants) | 154 | 153 | 84 | 70 | 83 | 70
percentage of participants | 26.0 | 41.8 | 29.8 | 21.4 | 44.6 | 38.6
Statistical Analysis 1: Comparison: Placebo vs Adalimumab Every Week (EW); Test type: Superiority or Other; p = 0.003, Cochran-Mantel-Haenszel — P-value adjusted for baseline Hurley Stage; Adjusted mean difference = 15.9, 95% CI 2-sided [5.3 to 26.5]
Statistical Analysis 2: Comparison: Placebo - Baseline Hurley Stage II vs Adalimumab Every Week (EW) - Baseline Hurley Stage II; Test type: Superiority or Other; p = 0.048, Chi-squared; Mean Difference (Final Values) = 14.8, 95% CI 2-sided [0.3 to 29.3]
Statistical Analysis 3: Comparison: Placebo - Baseline Hurley Stage III vs Adalimumab Every Week (ew) - Baseline Hurley Stage III; Test type: Superiority or Other; p = 0.027, Chi-squared; Mean Difference (Final Values) = 17.1, 95% CI 2-sided [2.2 to 32.1]

2. Secondary Outcome: Percentage of Participants With Baseline Hurley Stage II Who Achieved Abscess and Inflammatory Nodule (AN) Count of 0, 1, or 2 at Week 12
Description: The percentage of participants with AN counts lowered to 0, 1, or 2 at Week 12 among participants with Hurley Stage II at Baseline. NRI: Participants with missing data were considered non-responders.
Time Frame: Baseline (Week 0) up to Week 12
Population: Participants in the ITT population with baseline Hurley Stage II
Measure: Number; unit: percentage of participants
Arm/Group | Placebo - Baseline Hurley Stage II | Adalimumab Every Week (EW) - Baseline Hurley Stage II
Number analyzed (Participants) | 84 | 83
percentage of participants | 28.6 | 28.9
Statistical Analysis 1: Comparison: Placebo - Baseline Hurley Stage II vs Adalimumab Every Week (EW) - Baseline Hurley Stage II; Secondary end points 1 (AN 0/1/2 counts), 2 (NRS30), and 3 (modified Sartorius score) were ranked analyses; Test type: Superiority or Other; p = 0.961, Chi-squared; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-13.4 to 14.1]

3. Secondary Outcome: Percentage of Participants Achieving At Least 30% Reduction and At Least 1 Unit Reduction From Baseline in Patient's Global Assessment of Skin Pain (NRS30) - At Worst at Week 12 Among Participants With Baseline Skin Pain NRS ≥ 3
Description: The Patient's Global Assessment of Skin Pain Numeric Rating Scale (NRS) was used to assess the worst skin pain and the average skin pain due to HS. Ratings for the 2 items range from 0 (no skin pain) to 10 (skin pain as bad as you can imagine). The assessments were completed on a daily diary by participants before they went to bed and responded to the items based on a recall period of the "last 24 hours." The percentage of participants who achieved at least 30% reduction and at least 1 unit reduction from Baseline in the Patient's Global Assessment of Skin Pain (NRS30) - at worst at Week 12 among participants with Baseline NRS ≥ 3 are presented. Weekly averages of daily assessments were analyzed. NRI: Participants with missing data were considered non-responders.
Time Frame: Baseline (Week 0) up to Week 12
Population: Participants in the ITT population with baseline NRS at Worst ≥ 3
Measure: Number; unit: percentage of participants
Groups:
- Placebo - Baseline NRS at Worst ≥ 3: Participants with baseline NRS ≥ 3 randomized to receive placebo every week (ew) for 12 weeks.
- Adalimumab Every Week (EW) - Baseline NRS at Worst ≥ 3: Participants with baseline NRS ≥ 3 randomized to receive adalimumab ew 160 mg at Week 12, 80 mg at Week 14, and 40 mg ew from Week 16 to 35 (up to 24 weeks).
Arm/Group | Placebo - Baseline NRS at Worst ≥ 3 | Adalimumab Every Week (EW) - Baseline NRS at Worst ≥ 3
Number analyzed (Participants) | 109 | 122
percentage of participants | 24.8 | 27.9
Statistical Analysis 1: Comparison: Placebo - Baseline NRS at Worst ≥ 3 vs Adalimumab Every Week (EW) - Baseline NRS at Worst ≥ 3; Secondary end points 1 (AN 0/1/2 counts), 2 (NRS30), and 3 (modified Sartorius score) were ranked analyses; Test type: Superiority or Other; p = 0.628, Cochran-Mantel-Haenszel — P-value adjusted for baseline Hurley Stage; Adjusted mean difference = 2.8, 95% CI 2-sided [-8.6 to 14.2]

4. Secondary Outcome: Change From Baseline to Week 12 in Modified Sartorius Score
Description: The Sartorius Scale is used to quantify the severity of HS. Points are awarded for 12 body areas (left and right axillae, left and right sub/inframammary areas, intermammary area, left and right buttocks, left and right inguino-crural folds, perianal area, perineal area, and other): points were awarded for nodules (2 points for each); abscesses (4 points); fistulas (4 points); scars (1 point); other findings (1 point); and longest distance between two lesions (2-6 points, 0 if no lesions); and if lesions are separated by normal skin (yes-0 points; No-6 points). The total Sartorius score is the sum of the 12 regional scores. Last Observation Carried Forward (LOCF): The last completed evaluation from the previous visit within the particular period for efficacy measures was carried forward to impute missing data at later visits in the same period. Baseline efficacy evaluations were not carried forward.
Time Frame: Baseline (Week 0) and Week 12
Population: Participants in the ITT population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Adalimumab Every Week (EW)
Number analyzed (Participants) | 151 | 153
units on a scale | -15.7 (4) | -24.4 (3.97)
Statistical Analysis 1: Comparison: Placebo vs Adalimumab Every Week (EW); Secondary end points 1 (AN 0/1/2 counts), 2 (NRS30), and 3 (modified Sartorius score) were ranked analyses; Test type: Superiority or Other; p = 0.124, ANCOVA; P-value calculated from ANCOVA with stratum, baseline, and treatment as covariates; LS mean difference = -8.7, 95% CI 2-sided [-19.7 to 2.4]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from first dose of study drug until 70 days following last dose of study drug (46 weeks); Serious Adverse Events were collected from the time that informed consent was obtained (up to 50 weeks).
Description: Adverse Events with onset in Period 1 were collected from first dose of study drug until prior to the first dose in Period 2, or up to 70 days following last dose of study drug if the participant discontinued during Period 1.
Groups:
- Placebo (Period 1): Placebo for 12 weeks
- Adalimumab EW (Period 1): Adalimumab every week (ew) for 12 weeks (160 mg at Week 0; 80 mg at Week 2; and 40 mg ew from Week 4 to Week 12).
- Placebo/Adalimumab EW (Period 2): Participants randomized to receive placebo in Period 1 were re-randomized to receive adalimumab 160 mg at Week 12, 80 mg at Week 14, and 40 mg every week (ew) from Week 16 to Week 35 in Period 2 (up to 24 weeks).
- Adalimumab EW/Placebo (Period 2): Participants randomized to receive adalimumab every week (ew) in Period 1 were re-randomized to receive placebo ew from Week 12 to Week 35 in Period 2 (up to 24 weeks).
- Adalimumab EW/Adalimumab EOW (Period 2): Participants randomized to receive adalimumab every week (ew) in Period 1 were re-randomized to receive adalimumab 40 mg every other week (eow) from Week 12 to Week 35 in Period 2; placebo injections were administered eow from Week 13 to Week 35 (up to 24 weeks).
- Adalimumab EW/Adalimumab EW (Period 2): Participants randomized to receive adalimumab every week (ew) in Period 1 were re-randomized to receive 40 mg adalimumab ew from Week 12 to Week 35 in Period 2 (up to 24 weeks).
Arm/Group | Placebo (Period 1) | Adalimumab EW (Period 1) | Placebo/Adalimumab EW (Period 2) | Adalimumab EW/Placebo (Period 2) | Adalimumab EW/Adalimumab EOW (Period 2) | Adalimumab EW/Adalimumab EW (Period 2)
Serious Adverse Events (participants affected / at risk) | 5/152 | 3/153 | 5/145 | 2/49 | 3/48 | 1/48
Other Adverse Events (participants affected / at risk) | 81/152 | 64/153 | 68/145 | 30/49 | 24/48 | 28/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Period 1) (N=152) | Adalimumab EW (Period 1) (N=153) | Placebo/Adalimumab EW (Period 2) (N=145) | Adalimumab EW/Placebo (Period 2) (N=49) | Adalimumab EW/Adalimumab EOW (Period 2) (N=48) | Adalimumab EW/Adalimumab EW (Period 2) (N=48)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
EFFUSION (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
PNEUMONIA (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
PYELONEPHRITIS (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
HEPATITIS A ANTIBODY POSITIVE (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
LIVER FUNCTION TEST ABNORMAL (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
INTERVERTEBRAL DISC CALCIFICATION (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
TENDONITIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
INVASIVE DUCTAL BREAST CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
ECTOPIC PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 1
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
HIDRADENITIS (Skin and subcutaneous tissue disorders) | 3 | 1 | 2 | 2 | 2 | 0
ABORTION INDUCED (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Period 1) (N=152) | Adalimumab EW (Period 1) (N=153) | Placebo/Adalimumab EW (Period 2) (N=145) | Adalimumab EW/Placebo (Period 2) (N=49) | Adalimumab EW/Adalimumab EOW (Period 2) (N=48) | Adalimumab EW/Adalimumab EW (Period 2) (N=48)
ANAEMIA (Blood and lymphatic system disorders) | 1 | 1 | 1 | 1 | 0 | 2
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 | 0 | 2 | 1 | 0 | 0
NEUTROPHILIA (Blood and lymphatic system disorders) | 1 | 0 | 1 | 1 | 0 | 0
VERTIGO (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
HYPOTHYROIDISM (Endocrine disorders) | 0 | 0 | 1 | 0 | 1 | 0
BLEPHARITIS (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
EYELID OEDEMA (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
MEIBOMIAN GLAND DYSFUNCTION (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
VISUAL IMPAIRMENT (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 3 | 1 | 1 | 2 | 0 | 0
CONSTIPATION (Gastrointestinal disorders) | 2 | 1 | 1 | 0 | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 2 | 3 | 3 | 1 | 0 | 1
DRY MOUTH (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
GASTRITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
LIP SWELLING (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
NAUSEA (Gastrointestinal disorders) | 4 | 3 | 6 | 0 | 0 | 2
TOOTHACHE (Gastrointestinal disorders) | 1 | 0 | 2 | 1 | 0 | 0
VOMITING (Gastrointestinal disorders) | 2 | 1 | 1 | 1 | 1 | 1
CHILLS (General disorders) | 1 | 0 | 0 | 0 | 0 | 1
FATIGUE (General disorders) | 4 | 3 | 2 | 0 | 0 | 0
INJECTION SITE BRUISING (General disorders) | 0 | 1 | 1 | 1 | 0 | 0
INJECTION SITE ERYTHEMA (General disorders) | 0 | 1 | 6 | 0 | 0 | 0
INJECTION SITE PRURITUS (General disorders) | 0 | 1 | 3 | 0 | 0 | 1
LOCAL SWELLING (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
NON-CARDIAC CHEST PAIN (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
PYREXIA (General disorders) | 3 | 1 | 2 | 0 | 3 | 2
XEROSIS (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
CHOLELITHIASIS (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
HYPERSENSITIVITY (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0
BODY TINEA (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
BRONCHITIS (Infections and infestations) | 2 | 0 | 3 | 0 | 1 | 0
CELLULITIS (Infections and infestations) | 2 | 2 | 0 | 1 | 0 | 0
CYTOLYTIC VAGINOSIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
EAR INFECTION (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
FOLLICULITIS (Infections and infestations) | 1 | 0 | 2 | 0 | 1 | 2
IMPETIGO (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
INFLUENZA (Infections and infestations) | 3 | 2 | 3 | 0 | 0 | 1
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 0 | 0 | 1 | 1 | 0
MEASLES (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
NASOPHARYNGITIS (Infections and infestations) | 16 | 9 | 11 | 9 | 1 | 3
ORAL HERPES (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 0
OTITIS MEDIA (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
PHARYNGITIS (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 1 | 1 | 2 | 1 | 0 | 0
PNEUMONIA (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 0
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
RASH PUSTULAR (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
RHINITIS (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 0
SINUSITIS (Infections and infestations) | 1 | 3 | 4 | 1 | 0 | 2
SKIN CANDIDA (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 0
TINEA INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
TONSILLITIS (Infections and infestations) | 1 | 1 | 2 | 1 | 1 | 0
TRACHEITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 | 5 | 5 | 2 | 3 | 4
URINARY TRACT INFECTION (Infections and infestations) | 3 | 5 | 4 | 1 | 2 | 2
CONTUSION (Injury, poisoning and procedural complications) | 2 | 0 | 2 | 1 | 0 | 0
EXCORIATION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
FALL (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0 | 0 | 1
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0
SKIN INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 0 | 2 | 2 | 0 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 1 | 2 | 1 | 0 | 0
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
BLOOD GLUCOSE INCREASED (Investigations) | 0 | 0 | 1 | 0 | 1 | 0
BLOOD TRIGLYCERIDES INCREASED (Investigations) | 1 | 0 | 0 | 1 | 0 | 0
C-REACTIVE PROTEIN INCREASED (Investigations) | 3 | 3 | 2 | 1 | 0 | 0
WEIGHT DECREASED (Investigations) | 0 | 2 | 0 | 0 | 0 | 2
WEIGHT INCREASED (Investigations) | 3 | 3 | 2 | 0 | 0 | 1
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1
HYPERLIPIDAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 | 3 | 1 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 4 | 3 | 1 | 1 | 0 | 1
INTERVERTEBRAL DISC DEGENERATION (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3 | 1 | 0 | 0
DIZZINESS (Nervous system disorders) | 2 | 4 | 1 | 1 | 2 | 0
HEADACHE (Nervous system disorders) | 15 | 14 | 9 | 4 | 3 | 2
LETHARGY (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1
NERVE COMPRESSION (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
PARAESTHESIA (Nervous system disorders) | 1 | 0 | 1 | 1 | 0 | 0
SINUS HEADACHE (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1
SYNCOPE (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
DEPRESSION (Psychiatric disorders) | 0 | 3 | 2 | 1 | 0 | 0
INSOMNIA (Psychiatric disorders) | 1 | 1 | 1 | 0 | 1 | 2
DYSURIA (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
HAEMATURIA (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 2 | 0 | 1 | 2
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 3 | 1 | 0 | 0
RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 1
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0 | 1
SNEEZING (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
ACNE CYSTIC (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
DERMAL CYST (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 1 | 0 | 0
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 3 | 0
DERMATITIS PAPILLARIS CAPILLITII (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
DERMATITIS PSORIASIFORM (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 1
ECZEMA (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 0 | 0
ECZEMA ASTEATOTIC (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
HIDRADENITIS (Skin and subcutaneous tissue disorders) | 17 | 13 | 14 | 8 | 7 | 2
INTERTRIGO (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 1 | 0 | 2
KELOID SCAR (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
HYPERTENSION (Vascular disorders) | 3 | 1 | 2 | 2 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.